CLINICAL TRIAL: NCT01940237
Title: A Pilot Trial of Interpersonal Psychotherapy for the Treatment of Depression in Patients With Prostate, Colorectal, Lung and Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6397
Record Dates: First submitted 2013-08-28; First posted 2013-09-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Depression; Pancreatic Cancer; Lung Cancer; Colon Cancer; Prostate Cancer
Keywords: Depression; Psychotherapy; Cancer; Pancreatic Cancer; Lung Cancer; Colon Cancer; Prostate Cancer
MeSH Terms: conditions — Depression; Pancreatic Neoplasms; Lung Neoplasms; Colonic Neoplasms; Prostatic Neoplasms; Neoplasms | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interpersonal Psychotherapy (IPT) (Experimental): Interpersonal psychotherapy (IPT) is a brief, manualized therapy that has shown efficacy in the treatment of major depressive disorder (MDD) in several controlled trials. This study will test the efficacy of IPT in a group of prostate, colorectal, lung and pancreatic cancer patients with a diagnosis of major depressive disorder.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Interpersonal psychotherapy in the treatment of major depressive disorder.

SUMMARY:
There is now overwhelming evidence documenting the efficacy of psychotherapy in the treatment of depression in the general population. Surprisingly, however, given the high prevalence of depression in cancer patients, there are very few studies on the efficacy of psychotherapy in this population. Published studies of psychotherapy in cancer patients generally include patients with high heterogeneity of psychiatric diagnosis and frequently include patients without a psychiatric diagnosis, with the aim of preventing the appearance of a psychiatric disorder. This heterogeneity complicates the interpretation of the efficacy and specificity of these interventions. Specifically, the efficacy of psychotherapy for major depression in patients with cancer is unknown.

DETAILED DESCRIPTION:
Interpersonal psychotherapy (IPT) is a brief, manualized therapy that has shown efficacy in the treatment of major depressive disorder (MDD) in several controlled trials. This study will test the efficacy of IPT in a group of prostate, colorectal, lung and pancreatic cancer patients with a diagnosis of major depressive disorder.

We will test the efficacy of IPT using a variety of outcome measures at different time points of the treatment. Those scales will evaluate the patient's depressive symptoms, psychosocial functioning and quality of life. Patients that are deemed eligible for the study will have IPT for twelve weeks. Patients will receive twelve 50-minute sessions over 16 weeks. To facilitate access to treatment, sessions 1,2,3,4, 8 and 12 will be in person, while all others will in be person or over the telephone according to the patient's choice. Sessions will be audiotaped and periodically reviewed by experienced supervisors to assess therapist's adherence to IPT technique. This taping will be optional and is covered in a separate consent form. This pilot study is to prove feasibility and acceptability of IPT in this population and to show preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* A primary psychiatric diagnosis of Major Depressive Disorder as defined by DSM-IV
* Diagnosis of prostate, colorectal, lung or pancreatic cancer (stage 1-4)
* A score of 16 or above in the 17-item HAM-D (Hamilton depression scale)
* Male or female ages 18-75.
* Ability to give consent
* English and/ or Spanish Speaking

Exclusion Criteria:

* Lifetime history of psychosis or bipolar disorder
* History of substance abuse or dependence in the three months prior to the study.
* Current suicide risk.
* Patients who have ever failed IPT in the context of cancer.
* Patients who are receiving effective medication for depression
* Patients with T3, T4 and THS abnormal values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Scale (HAMD-17) | baseline, and every fourth week till week 12.
  10 to 15 minutes of mood assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Blanco, MD, PhD, Principal Investigator — NYSPI - Columbia University Medical Center
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States